CLINICAL TRIAL: NCT01304095
Title: Ranolazine, Ethnicity and the Metabolic Syndrome - REMS Study
Brief Title: Ranolazine, Ethnicity and the Metabolic Syndrome
Acronym: REMS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Atlanta Heart Specialists, LLC (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Principal Investigator, Narendra Singh, MD, Director, Clinical Research-AHS, Atlanta Heart Specialists, LLC
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AHS-REMS-001
Record Dates: First submitted 2011-02-16; First posted 2011-02-25 (Estimated); Last update posted 2013-07-11 (Estimated); Status verified 2013-07

CONDITIONS: Coronary Artery Disease; Angina; Metabolic Syndrome
Keywords: Coronary Artery Disease, Angina, Metabolic Syndrome
MeSH Terms: conditions — Coronary Artery Disease; Angina Pectoris; Metabolic Syndrome | interventions — Ranolazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ranolazine (Active Comparator): Ranolazine in addition to standard of care medical therapy
  Interventions: Drug: Ranolazine
- Standard of Care (No Intervention)

INTERVENTIONS:
Drug: Ranolazine — Patients in the ranolazine arm would start with 500 mg po BID of ranolazine and be force titrated to 1gm po BID after 2 weeks. Down-titration would only be allowed for side effects. This would be on top of all standard medical therapy.
  Other Names: Ranexa
  Arms: Ranolazine

SUMMARY:
The purpose of this study is to measure the effect of ranolazine on ETT (exercise treadmill test) exercise duration in four ethnic subgroups with established coronary artery disease and risk factor(s) for the metabolic syndrome: Caucasian, African American, Southeast Asian and East Indian.

DETAILED DESCRIPTION:
Studies have shown that various ethnic subgroups are at differential risk for both the development and progression of coronary artery disease. The East Indian population is one of the highest risk populations for coronary artery disease. Much of this increased risk is driven by the development and progression of diabetes.

Recent studies have shown that ranolazine has a favorable effect on glycemic control. In addition, it is an effective antianginal and antiarrhythmic agent.

The investigators propose a pilot study look at the safety, tolerability and efficacy of this agent in patients with established coronary artery disease (CAD) and risk factors for the metabolic syndrome from various ethnic backgrounds. In particular the investigators will focus on the Caucasian, African American, Southeast Asian and East Indian population.

ELIGIBILITY:
Inclusion Criteria:

1. Evidence of stable Coronary Artery Disease

   * MI > 30 days prior to enrollment
   * PCI > 30 days prior to enrollment
   * CABG > 30 days prior to enrollment
   * Angiography showing > 50% stenosis in a major vessel, branch or bypass graft > 30 days prior to enrollment
2. Metabolic Syndrome as evidenced by at least one of the following risk factors:

   * Abdominal Obesity (elevated waist circumference)

     * Men - waist circumference ≥ 40 inches (102 cm) Asians/Asian Americans ≥ 35.5 inches (90 cm)
     * Women - waist circumference ≥ 35 inches (88 cm) Asians/Asian Americans ≥ 31.5 inches (80 cm)
   * Atherogenic dyslipidemia (either one or both)

     * Triglycerides ≥ 150 mg/dL
     * Reduced HDL Men - HDL ≤ 40 mg/dL Women - HDL ≤ 50 mg/dL
   * Elevated Blood Pressure (equal to or greater than 130/85)
   * Elevated fasting glucose (equal to or greater than 100 mg/dL)
3. Symptoms of angina or a suspected angina equivalent (upper body chest pain, shortness of breath, fatigue)
4. Patient able to perform an exercise treadmill test (ETT)
5. Written informed consent
6. Age > 18 years old

Exclusion Criteria:

* Unstable coronary artery disease or revascularization within 30 days of enrollment.
* Patients who have a prolonged QTc interval (>500ms)
* Patients who have known severe liver disease
* Current or planned co-administration of strong CYP3A inhibitors (eg, ketoconazole, itraconazole, clarithromycin, nefazodone, nelfinavir, ritonavir, indinavir, and saquinavir) OR CYP3A inducers (eg, rifampin, rifabutin, rifapentine, Phenobarbital, phenytoin, carbamazepine, and St. John's Wort) OR moderate CYP3A inhibitors (eg, diltiazem, verapamil, aprepitant, erythromycin, fluconazole, and grapefruit juice or grapefruit-containing products)
* Patients who are pregnant or lactating
* Patients who are likely to be noncompliant with study procedures
* Patients currently in a study, or within 30 days of participating in a study, of an investigational drug or device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2011-01; Primary Completion 2013-07 (Actual); Study Completion 2013-11 (Estimated)

PRIMARY OUTCOMES:
Exercise Duration | change from baseline to 6 months
  To measure the effect of ranolazine on ETT (exercise treadmill test) exercise duration in four ethnic subgroups with established coronary artery disease and risk factor(s) for the metabolic syndrome: Caucasian, African American, Southeast Asian and East Indian.

SECONDARY OUTCOMES:
fasting glucose | change from baseline to 6 months
  To measure the effect ranolazine has on fasting blood glucose.
Angina | change from baseline to 6 months
  To look at the effect of ranolazine on anginal episodes using the Seattle Angina Questionnaire (SAQ).
Concomitant medications | change from baseline to 6 months
  To measure the impact of ranolazine on reducing concomitant medication therapy such as anti-arrhythmic agents, hypoglycemic agents, and nitrates.
lipid profile | change from baseline to 6 months
  To measure the effect ranolazine has on lipid profile.
HgbA1c | change from baseline to 6 months
  To measure the effect ranolazine has on hemoglobin A1c.

CONTACTS AND LOCATIONS:
Overall Officials: Narendra Singh, MD, Principal Investigator — Atlanta Heart Specialists, LLC
Locations (2):
- United States (2):
  - Atlanta Heart Specialist, LLC, Cumming, Georgia
  - Atlanta Heart Specialists, LLC, Tucker, Georgia